CLINICAL TRIAL: NCT05927883
Title: Efficacy of Indigenously Adapted Cognitive Behavioral Therapy for Reducing Gaming Addiction Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Ambreen Fatima, Principal Investigator, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-276182-002
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): Adolescents who scored high on IGD-SF-9. The group will be given IACBTGA
  Interventions: Behavioral: Indigenously Adapted Cognitive Behavioral Therapy
- Intervention group with Parental Psycho-education (Active Comparator): Adolescents who scored high on IGD-SF-9, parents of adolescents will also be added in intervention and CBT based psycho-education will be provided to parents and adolescents will be provided IACBTGA.
  Interventions: Behavioral: Indigenously Adapted Cognitive Behavioral Therapy
- Control (No Intervention): This group will not be given no intervention

INTERVENTIONS:
Behavioral: Indigenously Adapted Cognitive Behavioral Therapy — IACBTGA will be comprised of 8 weekly sessions. Cognitive and behavioral strategies will be provided in sessions
  Arms: Intervention group; Intervention group with Parental Psycho-education

SUMMARY:
Research evidence identified internet gaming as an emerging problem in youth across the globe and a lot of interventions are being used for managing gaming and associated psychological problems considering cultural aspects. Therefore, the present study aims at investigating the efficacy of Indigenously adapted cognitive behavior therapy for internet gaming addiction among Pakistani Youth. For this purpose, adolescents enrolled in 8th-12th grades in elementary and higher secondary schools in twin cities of Pakistan. Adolescents who scored high on Internet gaming disorder in screening will be included in the study and further detailed investigation will be completed by administering semi-structured Clinical Interviews, Coping inventory, self-control, and social connectedness. Participants will be divided into 2 groups i.e. experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents ranging from 13 - 19 years (WHO, 2013) enrolled in an educational institute in the vicinity of the Federal capital area
2. Playing Internet offline/online games.
3. Excessive users who play more than 5-8 hours per day,40 hours per week will be included.
4. Playing games for at least the past year.
5. No history of major illness or any other psychological disorder.

Exclusion Criteria:

1. Diagnosed prior for any mental or psychological disorder.
2. Receiving any psychotherapy or medication for any particular disorder

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Internet Gaming Disorder Scale - short form | 1 year
  Screening tool for internet gaming addiction based on DSM-5 criteria; Minimum score will be 9 and maximum score will be 45. Cutoff score is 25.

SECONDARY OUTCOMES:
Brief Self-Control Scale | 1 year
  The scale measures an individual's self-control. Minimum score will be 13 and maximum score will be 65. Higher score indicate low self control

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria University, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No